CLINICAL TRIAL: NCT06631547
Title: Effect of Progesterone Administration on Severely Head Injured Patients: Hospital Based Study
Brief Title: Effect of Progesterone Administration on Severely Head Injured Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Islam Abd El Aal Helmy, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pgs in head trauma
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Severe Head Trauma
MeSH Terms: conditions — Craniocerebral Trauma | interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Intramuscular injection of progesterone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients with main lines of management without progesterone (Placebo Comparator): patients with main lines of management without progesterone
  Interventions: Drug: The usual head trauma care
- Patients taking progesterone plus the main lines of management of traumatic brain injury (Active Comparator): taking progesterone IM 1mg/kg twice for 5 days plus the main lines of management of traumatic brain injury
  Interventions: Drug: Progesterone; Drug: The usual head trauma care

INTERVENTIONS:
Drug: Progesterone — Hormonal treatment
  Arms: Patients taking progesterone plus the main lines of management of traumatic brain injury
Drug: The usual head trauma care — the basic treatment

SUMMARY:
To investigate the effectiveness of progesterone as a neuroprotective in patients severe traumatic brain injury in clinical outcome

ELIGIBILITY:
Inclusion Criteria:patients with severe traumatic head injury GCS ≤8 both sexes.

>16yrs,

-

Exclusion Criteria:

* -Tumor that may flare with progesterone.
* patients with spinal injuries with neurological deficits.
* severe chest trauma that causes shock and hypoxia.
* life-threatening systemic injuries that cause hemodynamic instability, cardiac arrest
* pegnancy

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Glasgow outcome scale GOS-E score | 1year
  as thhe following:1-indicates death 2-indicates a vegetative state, 3 or 4 indicates a severe disability, 5 or 6 indicates a moderate disability and 7 or 8 indicates a good recovery. (8, 9)
FIM score | 1 year
  is available measure of dependence in two subscales (motor and cognitive) (10) . Motor domains self care (eating, grooming, bathing, body upper dressing, body lower dressing, swallowing, moving to bed and chair, toileting

SECONDARY OUTCOMES:
mortality rate | 1 month
  death rate at 1 month
Duration of hospital stay | 1month
  Duration of hospital stay
Duration of mechanical ventilator | 1month
  Duration of mechanical ventilator
adverse events | 1 month
  adverse events
Gcs | 1 year
  Gcs

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brooks JC, Strauss DJ, Shavelle RM, Paculdo DR, Hammond FM, Harrison-Felix CL. Long-term disability and survival in traumatic brain injury: results from the National Institute on Disability and Rehabilitation Research Model Systems. Arch Phys Med Rehabil. 2013 Nov;94(11):2203-9. doi: 10.1016/j.apmr.2013.07.005. Epub 2013 Jul 16. PMID 23872079
- [Background] Wilson JT, Pettigrew LE, Teasdale GM. Structured interviews for the Glasgow Outcome Scale and the extended Glasgow Outcome Scale: guidelines for their use. J Neurotrauma. 1998 Aug;15(8):573-85. doi: 10.1089/neu.1998.15.573. PMID 9726257
- [Background] Jennett B, Bond M. Assessment of outcome after severe brain damage. Lancet. 1975 Mar 1;1(7905):480-4. doi: 10.1016/s0140-6736(75)92830-5. PMID 46957
- [Background] Sarkaki AR, Khaksari Haddad M, Soltani Z, Shahrokhi N, Mahmoodi M. Time- and dose-dependent neuroprotective effects of sex steroid hormones on inflammatory cytokines after a traumatic brain injury. J Neurotrauma. 2013 Jan 1;30(1):47-54. doi: 10.1089/neu.2010.1686. Epub 2012 Nov 16. PMID 21851230
- [Background] Finnie JW. Neuroinflammation: beneficial and detrimental effects after traumatic brain injury. Inflammopharmacology. 2013 Aug;21(4):309-20. doi: 10.1007/s10787-012-0164-2. Epub 2013 Jan 8. PMID 23296919
- [Background] VanLandingham JW, Cekic M, Cutler S, Hoffman SW, Stein DG. Neurosteroids reduce inflammation after TBI through CD55 induction. Neurosci Lett. 2007 Sep 25;425(2):94-8. doi: 10.1016/j.neulet.2007.08.045. Epub 2007 Aug 25. PMID 17826908
- [Background] Guennoun R. Progesterone in the Brain: Hormone, Neurosteroid and Neuroprotectant. Int J Mol Sci. 2020 Jul 24;21(15):5271. doi: 10.3390/ijms21155271. PMID 32722286
- [Background] Werner C, Engelhard K. Pathophysiology of traumatic brain injury. Br J Anaesth. 2007 Jul;99(1):4-9. doi: 10.1093/bja/aem131. PMID 17573392
- [Background] Thapa K, Khan H, Singh TG, Kaur A. Traumatic Brain Injury: Mechanistic Insight on Pathophysiology and Potential Therapeutic Targets. J Mol Neurosci. 2021 Sep;71(9):1725-1742. doi: 10.1007/s12031-021-01841-7. Epub 2021 May 6. PMID 33956297
- [Background] Department Of Defense Washington DC. VA/DoD Clinical Practice Guideline for Management of Concussion/Mild Traumatic Brain Injury (mTBI). Ft. Belvoir: Defense Technical Information Center; 2009